CLINICAL TRIAL: NCT02555215
Title: A Multicenter Extension Study to Determine the Long-Term Safety and Efficacy of BG00012 in Pediatric Subjects With Relapsing-Remitting Multiple Sclerosis
Brief Title: Extension Study of BG00012 in Pediatric Subjects With Relapsing Remitting Multiple Sclerosis (RRMS)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 109MS311; 2015-003282-29 (EudraCT Number)
Record Dates: First submitted 2015-09-17; First posted 2015-09-21 (Estimated); Results first posted 2019-11-22 (Actual); Last update posted 2019-11-22 (Actual); Status verified 2019-11

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
Keywords: Pediatrics
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — Dimethyl Fumarate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- dimethyl fumarate (Experimental): Participants will receive 120 mg capsule(s) taken orally.
  Interventions: Drug: dimethyl fumarate

INTERVENTIONS:
Drug: dimethyl fumarate — administered orally
  Other Names: DMF; BG00012

SUMMARY:
The primary objective of the study is to evaluate the long-term safety of BG00012 in subjects who completed Study 109MS202 (NCT02410200). Secondary objectives are as follows: To evaluate the long-term efficacy of BG00012 and to describe the long-term Multiple Sclerosis (MS) outcomes in subjects who completed Study 109MS202 (NCT02410200).

ELIGIBILITY:
Key Inclusion Criteria:

* Ability of parents, legal guardians, and/or subjects to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use confidential health information in accordance with national and local subject privacy regulations. Subjects will provide assent in addition to the parental or guardian consent, as appropriate, per local regulations.
* Subjects who completed, as per protocol, the previous BG00012 clinical study 109MS202 (NCT02410200) and remain on BG00012 treatment.

Key Exclusion Criteria:

* Unwillingness or inability to comply with study requirements, including the presence of any condition (physical, mental, or social) that is likely to affect the subject's ability to comply with the protocol.
* Any significant changes in medical history occurring after enrollment in the parent Study 109MS202 (NCT02410200), including laboratory test abnormalities or current clinically significant conditions that in the opinion of the Investigator would have excluded the subject's participation from the parent study. The Investigator must re-review the subject's medical fitness for participation and consider any factors that would preclude treatment.
* Subjects from Study 109MS202 (NCT02410200) who could not tolerate study treatment.

NOTE: Other protocol defined inclusion/exclusion criteria may apply.

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2016-02-22 (Actual); Primary Completion 2018-09-24 (Actual); Study Completion 2018-09-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (12):
- Research Site, Loma Linda, California, United States
- Research Site, Ghent, Belgium
- Research Site, Sofia, Bulgaria
- Research Site, Hradec Králové, Czechia
- Germany (2):
  - Research Site, Munich, Bavaria
  - Research Site, Göttingen, Lower Saxony
- Research Site, Kuwait City, Kuwait
- Research Site, Riga, Latvia
- Research Site, Beirut, Lebanon
- Poland (2):
  - Research Site, Gdansk
  - Research Site, Poznan
- Research Site, Ankara, Turkey (Türkiye)

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dimethyl Fumarate
Started | 20
Completed | 17
Not Completed | 3
Not completed — Other | 1
Not completed — Investigator Decision | 2

BASELINE CHARACTERISTICS:
Arm/Group | Dimethyl Fumarate
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 14
  Between 18 and 65 years | 6
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.7 (1.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 7
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 1
  Black or African American | 0
  White | 5
  Not Reported Due to Confidentiality Regulations | 13
  Other | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence that does not necessarily have a causal relationship with treatment. An SAE is any untoward medical occurrence that at any dose: results in death; in the view of the Investigator, places the participant at immediate risk of death (a life-threatening event); requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; results in a congenital anomaly/birth defect; any other medically important event that, in the opinion of the Investigator, may jeopardize the participant or may require intervention to prevent one of the other outcomes listed in the definition above.
Time Frame: Baseline to Week 96
Population: The safety population was defined as all participants who received at least 1 dose of BG00012.
Measure: Number; unit: participants
Arm/Group | Dimethyl Fumarate
Number analyzed (Participants) | 20
participants
  AE | 18
  SAE | 2

2. Primary Outcome: Number of Participants Discontinuing Treatment Due to an Adverse Event
Description: An AE is any untoward medical occurrence that does not necessarily have a causal relationship with treatment.
Time Frame: Baseline to Week 96
Measure: Number; unit: participants
Arm/Group | Dimethyl Fumarate
Number analyzed (Participants) | 20
participants | 0

3. Secondary Outcome: Total Number of New or Newly Enlarging T2 Hyperintense Lesions From Week 16 to Week 24
Description: T2 hyperintense lesions were measured by MRI brain scans.
Time Frame: Week 16 to Week 24
Population: Participants who received at least 1 dose of BG00012 in this study and had an evaluation of the efficacy endpoint under analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Dimethyl Fumarate
Number analyzed (Participants) | 17
Participants
  0 lesions | 12
  1 lesion | 2
  2 lesions | 1
  3 lesions | 1
  4 lesions | 0
  5 or more lesions | 1

4. Secondary Outcome: Total Number of New or Newly Enlarging T2 Hyperintense Lesions From Week 64 to Week 72
Description: T2 hyperintense lesions were measured by MRI brain scans.
Time Frame: Week 64 to Week 72
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Dimethyl Fumarate
Number analyzed (Participants) | 10
Participants
  0 lesions | 8
  1 lesion | 1
  2 lesions | 1
  3 lesions | 0
  4 lesions | 0
  5 or more lesions | 0

5. Secondary Outcome: Average Annualized Relapse Rate (ARR)
Description: Relapses were defined as new or recurrent neurologic symptoms not associated with fever or infection, lasting at least 24 hours, and accompanied by new objective neurological findings upon examination by the Investigator. New or recurrent neurologic symptoms that evolved gradually over months were considered disability progression, not an acute relapse, and were not treated with steroids.
  The ARR was calculated as the total number of relapses that occurred during the previous 12 months and during the 120 weeks on treatment for participants in Study 109MS202 that continued into Study 109MS311, divided by the total number of person-years followed prior to the study and by the total number of person-years followed during the study, respectively.
Time Frame: Baseline to Week 96
Population: as for outcome 3
Measure: Number; unit: relapses per person-years
Arm/Group | Dimethyl Fumarate
Number analyzed (Participants) | 20
relapses per person-years | 0.1

6. Secondary Outcome: Percentage of Participants Experiencing One or More Relapses
Description: Relapses were defined as new or recurrent neurologic symptoms not associated with fever or infection, lasting at least 24 hours, and accompanied by new objective neurological findings upon examination by the Investigator. New or recurrent neurologic symptoms that evolved gradually over months were considered disability progression, not an acute relapse, and were not treated with steroids.
Time Frame: Baseline to Week 96
Measure: Number; unit: percentage of participants
Arm/Group | Dimethyl Fumarate
Number analyzed (Participants) | 20
percentage of participants | 10

7. Secondary Outcome: Change From Baseline in the Degree of Disability
Description: The Expanded Disability Status Scale (EDSS) measures disability status on a scale ranging from 0 to 10, with higher scores indicating more disability. Scoring is based on measures of impairment in eight functional systems on examination by a neurologist.
Time Frame: Baseline to Week 96
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dimethyl Fumarate
Number analyzed (Participants) | 20
score on a scale
  Baseline | 1.00 (1.026)
  Change from Baseline at Week 12: number analyzed (Participants) | 13
  Change from Baseline at Week 12 | 0.15 (0.718)
  Change from Baseline at Week 24: number analyzed (Participants) | 14
  Change from Baseline at Week 24 | 0.29 (0.508)
  Change from Baseline at Week 36: number analyzed (Participants) | 13
  Change from Baseline at Week 36 | 0.27 (0.832)
  Change from Baseline at Week 48: number analyzed (Participants) | 9
  Change from Baseline at Week 48 | 0.50 (0.791)
  Change from Baseline at Week 72: number analyzed (Participants) | 12
  Change from Baseline at Week 72 | 0.71 (1.010)
  Change from Baseline at Week 96: number analyzed (Participants) | 12
  Change from Baseline at Week 96 | 0.21 (0.964)

8. Secondary Outcome: Number of Participants Experiencing Disability Progression
Description: Measured by at least a 1.0-point increase on the EDSS from baseline EDSS ≥1.0 that is sustained for 24 weeks, or at least a 1.5-point increase on the EDSS from baseline EDSS = 0 that is sustained for 24 weeks.
Time Frame: Baseline to Week 96
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Dimethyl Fumarate
Number analyzed (Participants) | 20
Participants | 3

ADVERSE EVENTS:
Time Frame: Baseline to Week 96
Groups:
- BG00012: Participants will receive 120 mg capsule(s) taken orally.
Arm/Group | BG00012
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 2/20
Other Adverse Events (participants affected / at risk) | 18/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BG00012 (N=20)
Abdominal pain (Gastrointestinal disorders) | 1
Multiple sclerosis relapse (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BG00012 (N=20)
Vertigo (Ear and labyrinth disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 3
Abdominal pain upper (Gastrointestinal disorders) | 2
Fatigue (General disorders) | 2
Gastroenteritis (Infections and infestations) | 2
Nasopharyngitis (Infections and infestations) | 2
Pharyngitis (Infections and infestations) | 2
Upper respiratory tract infection (Infections and infestations) | 3
Viral upper respiratory tract infection (Infections and infestations) | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2
Headache (Nervous system disorders) | 3
Hypoaesthesia (Nervous system disorders) | 2
Multiple sclerosis relapse (Nervous system disorders) | 4
Dysmenorrhoea (Reproductive system and breast disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2
Acne (Skin and subcutaneous tissue disorders) | 2
Flushing (Vascular disorders) | 5
Wolff-parkinson-white syndrome (Cardiac disorders) | 1
Eye irritation (Eye disorders) | 1
Vision blurred (Eye disorders) | 1
Abdominal discomfort (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Dry mouth (Gastrointestinal disorders) | 1
Mouth ulceration (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Influenza like illness (General disorders) | 1
Dust allergy (Immune system disorders) | 1
Seasonal allergy (Immune system disorders) | 1
Smoke sensitivity (Immune system disorders) | 1
Cystitis (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Mastoiditis (Infections and infestations) | 1
Respiratory tract infection viral (Infections and infestations) | 1
Root canal infection (Infections and infestations) | 1
Salpingo-oophoritis (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Tonsillitis (Infections and infestations) | 1
Burns second degree (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 1
Ligament sprain (Injury, poisoning and procedural complications) | 1
Limb injury (Injury, poisoning and procedural complications) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Demyelination (Nervous system disorders) | 1
Migraine (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 1
Presyncope (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Irritability (Psychiatric disorders) | 1
Somatic symptom disorder (Psychiatric disorders) | 1
Dysuria (Renal and urinary disorders) | 1
Hypertonic bladder (Renal and urinary disorders) | 1
Micturition urgency (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Menstruation irregular (Reproductive system and breast disorders) | 1
Ovarian cyst (Reproductive system and breast disorders) | 1
Uterine inflammation (Reproductive system and breast disorders) | 1
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 1
Paranasal cyst (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Alopecia areata (Skin and subcutaneous tissue disorders) | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for noncommercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.

DOCUMENTS (2):
  • Study Protocol (2018-04-24): https://cdn.clinicaltrials.gov/large-docs/15/NCT02555215/Prot_000.pdf
  • Statistical Analysis Plan (2018-07-09): https://cdn.clinicaltrials.gov/large-docs/15/NCT02555215/SAP_001.pdf